CLINICAL TRIAL: NCT04982757
Title: COVID-19 Compatible Accelerated TMS Therapy
Brief Title: Accelerated TMS for Depression and OCD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: The New Venture Fund / Foundation for OCD Research (Unknown); The Wellcome Leap Fund (Unknown); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20-10022827; UG3MH137656 (NIH)
Record Dates: First submitted 2021-07-17; First posted 2021-07-29 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Depression; OCD
Keywords: TMS
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receive rTMS targeting the DMPFC or the LPFC. The treatment course will be 10 sessions per day hourly for 5 days. Participants may have the option to be crossed over to receive rTMS targeting the opposite brain area, enabling us to test whether participants who do not respond well to one target might respond to stimulation of another target. The option to offer a second course of treatment will be based on clinical judgement and re-evaluation of the participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Depression - DMPFC target to (for non-responders) LPFC target (Experimental): Participants with treatment resistant depression will receive a 5-day course of rTMS delivered to the DMPFC. Participants may have the option to be crossed over to receive rTMS targeting the opposite brain area (LPFC), enabling us to test whether participants who do not respond well to one target might respond to stimulation of another target. The option to offer a second course of treatment will be based on clinical judgement and re-evaluation of the participant.
  Interventions: Device: MagVenture MagPro System with Brainsight neuronavigation device
- Depression - LPFC target to (for non-responders) DMPFC target (Active Comparator): Participants with treatment resistant depression will receive a 5-day course of rTMS delivered to the LPFC. Participants may have the option to be crossed over to receive rTMS targeting the opposite brain area (DMPFC), enabling us to test whether participants who do not respond well to one target might respond to stimulation of another target. The option to offer a second course of treatment will be based on clinical judgement and re-evaluation of the participant.
  Interventions: Device: MagVenture MagPro System with Brainsight neuronavigation device
- OCD - DMPFC target to (for non-responders) LPFC target (Experimental): Participants with OCD will receive a 5-day course of rTMS delivered to the DMPFC.Participants may have the option to be crossed over to receive rTMS targeting the opposite brain area (LPFC), enabling us to test whether participants who do not respond well to one target might respond to stimulation of another target. The option to offer a second course of treatment will be based on clinical judgement and re-evaluation of the participant.
  Interventions: Device: MagVenture MagPro System with Brainsight neuronavigation device
- OCD - LPFC target to (for non-responders) DMPFC target (Active Comparator): Participants with OCD will receive a 5-day course of rTMS delivered to the LPFC. Participants may have the option to be crossed over to receive rTMS targeting the opposite brain area (DMPFC), enabling us to test whether participants who do not respond well to one target might respond to stimulation of another target. The option to offer a second course of treatment will be based on clinical judgement and re-evaluation of the participant.
  Interventions: Device: MagVenture MagPro System with Brainsight neuronavigation device

INTERVENTIONS:
Device: MagVenture MagPro System with Brainsight neuronavigation device — 10x daily sessions of 1200 pulses of theta-burst stimulation lasting approximately ten minutes.

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) is a FDA-approved treatment for depression and Obsessive Compulsive Disorder (OCD). The goal of the study is to learn how to optimize the treatment to improve symptoms of depression and OCD. This research project will test a new accelerated 5-day accelerated rTMS protocol for treating symptoms of depression and OCD.

A second goal of this study is to identify biomarkers of depression and OCD in the brain using functional magnetic resonance imaging (fMRI). This approach will predict who will benefit from TMS, determine the optimal treatment target, and improve treatment outcomes. Subjects will receive a clinical assessment of symptoms and an fMRI brain scan before and after each treatment course to measure the effect of treatment on symptom severity and on fMRI measures of functional connectivity.

Participants will be randomized to receive rTMS targeting either the lateral prefrontal cortex (LPFC) or the dorsomedial prefrontal cortex (DMPFC). Participants will complete a 5-day course of rTMS delivered hourly for 10 hours per day. Participants who show a partial response to treatment but not a full response will then receive a second 5-day course. Treatment non-responders will be crossed over to receive rTMS targeting the opposite brain area.

The primary hypothesis is that accelerated rTMS treatment will yield rapid improvement in symptoms for patients with depression and OCD in just 5 days, and that response rates can be further improved by adding a second 5-day treatment course.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depressive disorder OR obsessive-compulsive disorder (DSM-V criteria)
* Hamilton Depression Rating Scale score greater than or equal to 18 OR Yale-Brown Obsessive-Compulsive Scale score greater than or equal to 16
* Failed at least 1 prior trial of standard first-line treatment for depression or OCD per the modified Antidepressant Treatment History form and APA Practice Guidelines (e.g. serotonin reuptake inhibitor [SRI] or cognitive behavioral therapy with exposure and response prevention) OR had refused these treatments for individual reasons (e.g., cannot tolerate side effects, cannot tolerate exposure therapy, etc.).
* Off antidepressants OR on a stable dose of antidepressants for greater than or equal to four weeks with plans to remain on this stable dose during the study Note: Medications that are known to increase cortical excitability (e.g., buprorion, maprotiline, tricyclic antidepressants, classical antipsychotics) or to have an inhibitory effect on brain excitability (e.g., anticonvulsants, benzodiazepines, and atypical antipsychotics), or any other medications with relative hazard for use in TMS will be allowed upon review of medications and/or motor threshold determination by TMS specialist.
* Capacity to consent

Exclusion Criteria:

* Imminent risk of suicide (based on the CSSRS)
* Presence of primary psychiatric diagnoses other than OCD, MDD and/or co-morbid GAD (ex. PTSD, MDD with psychotic features, primary psychotic illness, Bipolar I or II)
* Evidence of cognitive impairment (MMSE score falling 1 SD below mean score for his/her age and education)
* Evidence of psychotic symptoms on diagnostic interview (interfering with capacity to consent)
* Have met criteria for any significant substance use disorder within the past 6 months
* Recent onset (within 8 weeks of screening) of psychotherapy
* Prior completion of this accelerated TMS treatment protocol during the current depressive episode
* Participated in any clinical trial with an investigational drug or device within the past 6 weeks prior to screening
* Evidence or history of significant neurological disorder including moderate-severe head trauma, stroke, Parkinson's disease or other movement disorder (except benign essential tremor), epilepsy
* History of seizures (except juvenile febrile seizures) or any condition/concurrent medication that could notably lower seizure threshold
* Presence of foreign metal bodies/implanted intracranial devices (MRI contraindication)
* Current pregnancy or planning to conceive during the study
* Abnormal bloodwork for electrolytes, thyroid or liver function

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-12-07 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Percent Change in Yale-Brown Obsessive Compulsive Scale (YBOCS) scores for participants with OCD | Baseline to Treatment End: Day 5, 10, 15, or 20 (depending on number of 5-day treatment courses administered)
  The YBOCS is a measure of obsessive compulsive symptoms is scored on a scale of 0 to 40, with 0 being no symptoms and 40 being extreme symptoms of OCD.
Change in Montgomery-Asberg Depression Rating Scale (MADRS) scores for participants with treatment resistant depression | Baseline to Treatment End: Day 5 or 10 (depending on number of 5-day treatment courses administered)
  The MADRS is a measure of depression symptoms and is scored on a scale of 0 to 60, with 0 being no depressive symptoms and 60 being severe depressive symptoms.

SECONDARY OUTCOMES:
Percent Change in Quick Inventory of Depressive Symptomatology (QIDS) scores for participants with OCD | Baseline to Treatment End: Day 5 or 10 (depending on number of 5-day treatment courses administered)
  The QIDS is a self-report measure of depression symptoms and is scored on a scale of 0 to 27, with 0 being no depressive symptoms and 27 being severe depressive symptoms.
Percent Change in Beck Depression Inventory (BDI) scores for participants with OCD | Baseline to Treatment End: Day 5 or 10 (depending on number of 5-day treatment courses administered)
  The BDI is a self-report measure of depression symptoms and is scored on a scale of 0 to 63, with 0 being no depressive symptoms and 63 being severe depressive symptoms.
Percent Change in Patient Health Questionnaire (PHQ-9) scores for participants with OCD | Baseline to Treatment End: Day 5 or 10 (depending on number of 5-day treatment courses administered)
  The PHQ-9 is a self-report measure of depression symptoms and is scored on a scale of 0 to 63, with 0 being no depressive symptoms and 63 being severe depressive symptoms.
Percent Change in Patient Health Questionnaire-9 (PHQ-9) scores for participants with OCD | Baseline to Treatment End: Day 5 or 10 (depending on number of 5-day treatment courses administered)
  The PHQ-9 is a self-report measure of depression symptoms and is scored on a scale of 0 to 63, with 0 being no depressive symptoms and 27 being severe depressive symptoms.
Percent Change in Beck Anxiety Inventory (BAI) scores for participants with OCD | Baseline to Treatment End: Day 5 or 10 (depending on number of 5-day treatment courses administered)
  The BAI is a self-report measure of anxiety symptoms and is scored on a scale of 0 to 63, with 0 being no anxiety symptoms and 63 being severe anxiety symptoms.
Percent Change in General Anxiety Disorder (GAD-7) scores for participants with OCD | Baseline to Treatment End: Day 5 or 10 (depending on number of 5-day treatment courses administered)
  The BAI is a self-report measure of anxiety symptoms and is scored on a scale of 0 to 21, with 0 being no anxiety symptoms and 21 being severe anxiety symptoms.
Percent Change in 17-item Hamilton Depression Rating Scale (HAM-D) scores for participants with treatment resistant depression | Baseline to Treatment End: Day 5 or 10 (depending on number of 5-day treatment courses administered)
  The HAM-D is a clinician-rated measure of depression symptoms and is scored on a scale of 0 to 52, with 0 being no anxiety symptoms and 21 being severe depression symptoms.
Percent Change in Beck Depression Inventory (BDI) scores for participants with treatment resistant depression | Baseline to Treatment End: Day 5 or 10 (depending on number of 5-day treatment courses administered)
  The BDI is a self-report measure of depression symptoms and is scored on a scale of 0 to 63, with 0 being no depressive symptoms and 63 being severe depressive symptoms.
Change in resting-state fMRI connectivity between the frontostriatal network and limbic network in participants with OCD | Baseline to Treatment End: Day 5 or 10 (depending on number of 5-day treatment courses administered)
  Change in resting state fMRI connectivity between the frontostriatal network and limbic network will be measured as a between-network correlational score of 0 to 1, with 0 low between-network connectivity and 1 being the highest possible between-network connectivity.
Change in resting-state fMRI connectivity between the frontostriatal network and limbic network in participants with treatment resistant depression | Baseline to Treatment End: Day 5 or 10 (depending on number of 5-day treatment courses administered)
  Change in resting state fMRI connectivity between the frontostriatal network and limbic network will be measured as a between-network correlational score of 0 to 1, with 0 low between-network connectivity and 1 being the highest possible between-network connectivity.

CONTACTS AND LOCATIONS:
Overall Officials: Conor Liston, MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual data collected during the trial will be available after deidentification upon request to the PI. Data to be shared include deidentified clinical assessment scores and MRI images.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Deidentified data will be available any time following publication of outcomes from this study, with no specified end date.
Access Criteria: Deidentified data will be shared with any researcher requesting access.